CLINICAL TRIAL: NCT03478891
Title: VRC 608: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-EBOMAB092-00-AB (MAb114), Administered Intravenously to Healthy Adults
Brief Title: Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-EBOMAB092-00-AB (MAb114), Administered Intravenously to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180069; 18-I-0069
Expanded Access: Available
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2018-10-11 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Healthy Adult Immune Responses to Vaccine
Keywords: Ebola Virus; Immune Response; Filovirus; Ebola Hemorrhagic Fever; First in Human
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — ansuvimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: 5 mg/kg IV (Experimental): Group 1 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 5 mg/kg.
  Interventions: Biological: VRC-EBOMAB092-00-AB (MAb114)
- Group 2: 25 mg/kg IV (Experimental): Group 2 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 25 mg/kg.
  Interventions: Biological: VRC-EBOMAB092-00-AB (MAb114)
- Group 3: 50 mg/kg IV (Experimental): Group 3 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 50 mg/kg.
  Interventions: Biological: VRC-EBOMAB092-00-AB (MAb114)

INTERVENTIONS:
Biological: VRC-EBOMAB092-00-AB (MAb114) — VRC-EBOMAB092-00-AB (MAb114) is a human immunoglobulin (IgG1) monoclonal antibody (MAb) targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP).

SUMMARY:
Background:

Ebola is a virus that has infected and killed people mostly in West Africa. There is no treatment or prevention for it, but several drugs are being studied. Researchers want to test the drug MAb114 in healthy people not exposed to Ebola to see whether it can be used for Ebola treatment in people who are infected in the future. This trial will not expose volunteers to the Ebola virus.

Objectives:

To see if MAb114 is safe and how a person's body responds to it.

Eligibility:

Healthy adults ages 18-60 who weigh 220.5 pounds or less

Design:

Participants will be screened under protocol NIH 11-I-0164 with:

* Medical history
* Physical exam
* Blood or urine tests

Participants will have a first 8- to10-hour visit. They will get MAb114 by IV infusion. For this, a thin tube will be placed in an arm vein. They may get an IV line in their other arm to collect blood. Blood will be taken many times before and after the infusion. Participants may have a urine test.

Participants will get a thermometer to check their temperature for 3 days after they get MAb114. They will record their highest temperature and any symptoms.

Participants will have about 14 more study visits over 6 months. At each visit, they will have blood taken and be checked for any health changes. They will talk about how they are feeling and if they have taken any medications.

At the end of the 6 months, participants may be invited to take part in another study for follow-up sample collection.

DETAILED DESCRIPTION:
VRC 608: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-EBOMAB092-00-AB (MAb114), Administered Intravenously to Healthy Adults

Study Design: VRC 608 is the first-in-human Phase I study to examine safety, tolerability and pharmacokinetics of the monoclonal antibody (MAb), VRC-EBOMAB092-00-AB (MAb114). MAb114 will be administered as a single dose. The hypotheses are: 1) MAb114 administration to healthy adults will be safe by the intravenous (IV) route; and 2) MAb114 will be detectable in human sera with a definable half-life. The primary objectives are to evaluate the safety and tolerability of MAb114 in healthy adults. Secondary objectives will evaluate the pharmacokinetics of MAb114 and the potential to detect an anti-drug antibody response to MAb114.

Product Description: MAb114 is a human IgG1 MAb targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP). It was developed by the VRC/NIAID/NIH and manufactured at Cook Pharmica LLC d.b.a. Catalent Indiana, LLC (Bloomington, IN) under current Good Manufacturing Practice (cGMP) regulations. MAb114 is supplied as a lyophilized product in a glass vial at 400 mg per vial with target overfill to 425 mg per vial.

Subjects: Up to 30 healthy adults, 18-60 years of age.

Study Plan: This is an open-label, dose-escalation study of MAb114 administered by IV infusion at dosages of 5, 25 and 50 mg/kg (Groups 1-3). Enrollment will begin with the lowest dose group. Following the first product administration in each group, the study team will wait at least 3 days before administering MAb114 to a second subject within the same group. Dose-escalation evaluations will occur to ensure the safety data support proceeding to the higher doses. Solicited reactogenicity following product administration will be evaluated using a 3-day diary. Assessment of safety will include clinical observation and monitoring of serum hematological and chemical parameters at defined timepoints throughout the study.

* Group 1: 3 subjects; 5 mg/kg IV
* Group 2: 5 subjects; 25 mg/kg IV
* Group 3: 10 subjects; 50 mg/kg IV
* Total* 18 subjects

  * A minimum of 18 subjects will be enrolled. Enrollment up to a total of 30 subjects is permitted if additional subjects are necessary for safety or pharmacokinetic (PK) evaluations.

Study Duration: Subjects will be followed for 24 weeks after the study product administration.

ELIGIBILITY:
INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

* Able and willing to complete the informed consent process.
* Available for clinical follow-up through the last study visit.
* 18 to 60 years of age.
* In good general health without clinically significant medical history.
* Willing to have blood samples collected, stored indefinitely, and used for research purposes.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* Physical examination without clinically significant findings within the 84 days prior to enrollment.
* Have screening laboratory values within 84 days prior to enrollment that meet the following criteria:

  * White Blood Cell (WBC) 2,500-12,000/mm^3
  * WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval
  * Platelets = 125,000 - 400,000/mm^3
  * Hemoglobin within institutional normal range or accompanied by the PI or designee approval
  * Creatinine less than or equal to 1.1 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) less than or equal to 1.25 x ULN
  * Negative for human immunodeficiency virus (HIV) infection by a Food and Drug Administration (FDA) approved method of detection
  * Negative for Hepatitis B core antibody (HBcAb) and Hepatitis C virus antibody (HCV Ab)
* Criteria applicable to women of childbearing potential:

  * If a woman is of reproductive potential and sexually active with a male partner, then she agrees to use an effective means of birth control from the time of study enrollment until the last study visit, or to be monogamous with a partner who has had a vasectomy.
  * Negative human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on day of enrollment and product administration.

EXCLUSION CRITERIA:

A volunteer will be excluded from study participation if one or more of the following conditions apply:

* Previous receipt of a licensed or investigational monoclonal antibody or Ebola vaccine.
* Weight >100 kg.
* Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study.
* Hypertension that is not well controlled.
* Woman who is breast-feeding, or planning to become pregnant during study participation.
* Receipt of any investigational study product within 28 days prior to enrollment.
* Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular (IM) injections or blood draws.
* Use of angiotensin-converting enzyme (ACE) inhibitors or other potential nephrotoxins.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corti D, Misasi J, Mulangu S, Stanley DA, Kanekiyo M, Wollen S, Ploquin A, Doria-Rose NA, Staupe RP, Bailey M, Shi W, Choe M, Marcus H, Thompson EA, Cagigi A, Silacci C, Fernandez-Rodriguez B, Perez L, Sallusto F, Vanzetta F, Agatic G, Cameroni E, Kisalu N, Gordon I, Ledgerwood JE, Mascola JR, Graham BS, Muyembe-Tamfun JJ, Trefry JC, Lanzavecchia A, Sullivan NJ. Protective monotherapy against lethal Ebola virus infection by a potently neutralizing antibody. Science. 2016 Mar 18;351(6279):1339-42. doi: 10.1126/science.aad5224. Epub 2016 Feb 25. PMID 26917593
- [Background] Misasi J, Gilman MS, Kanekiyo M, Gui M, Cagigi A, Mulangu S, Corti D, Ledgerwood JE, Lanzavecchia A, Cunningham J, Muyembe-Tamfun JJ, Baxa U, Graham BS, Xiang Y, Sullivan NJ, McLellan JS. Structural and molecular basis for Ebola virus neutralization by protective human antibodies. Science. 2016 Mar 18;351(6279):1343-6. doi: 10.1126/science.aad6117. Epub 2016 Feb 25. PMID 26917592
- [Result] Gaudinski MR, Coates EE, Novik L, Widge A, Houser KV, Burch E, Holman LA, Gordon IJ, Chen GL, Carter C, Nason M, Sitar S, Yamshchikov G, Berkowitz N, Andrews C, Vazquez S, Laurencot C, Misasi J, Arnold F, Carlton K, Lawlor H, Gall J, Bailer RT, McDermott A, Capparelli E, Koup RA, Mascola JR, Graham BS, Sullivan NJ, Ledgerwood JE; VRC 608 Study team. Safety, tolerability, pharmacokinetics, and immunogenicity of the therapeutic monoclonal antibody mAb114 targeting Ebola virus glycoprotein (VRC 608): an open-label phase 1 study. Lancet. 2019 Mar 2;393(10174):889-898. doi: 10.1016/S0140-6736(19)30036-4. Epub 2019 Jan 24. PMID 30686586
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-I-0069.html
- See also: NIH Press Release — https://www.nih.gov/news-events/news-releases/investigational-monoclonal-antibody-treat-ebola-safe-adults

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland
Period: Overall Study
Arm/Group | Group 1: 5 mg/kg IV | Group 2: 25 mg/kg IV | Group 3: 50 mg/kg IV
Started | 3 | 5 | 11
Received MAb114 | 3 | 5 | 10 (One Group 3 subject discontinued prior to MAb114 infusion due to inadequate venous access)
Completed | 2 | 5 | 8
Not Completed | 1 | 0 | 3
Not completed — Enrolled, but product never administered | 0 | 0 | 1
Not completed — Moved from area | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 5 mg/kg IV | Group 2: 25 mg/kg IV | Group 3: 50 mg/kg IV | Total
Number analyzed (Participants) | 3 | 5 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (7.4) | 36.4 (9.8) | 39.0 (13.9) | 38.4 (11.7)
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 0 | 1 | 4 | 5
  31-40 years | 2 | 2 | 2 | 6
  41-50 years | 1 | 2 | 1 | 4
  51-60 years | 0 | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 7 | 12
  Male | 2 | 1 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 4 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 2 | 5 | 7 | 14
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 11 | 19
Weight [Mean (Standard Deviation); unit: kg] | 88 (8.8) | 66.3 (12.6) | 73.5 (12.4) | 73.9 (13.4)
Education [Count of Participants; unit: Participants]
  College or University | 2 | 3 | 8 | 13
  Advanced Degree | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Infusion Reaction During Product Administration
Description: Possible infusion reaction symptoms: unusually tired/feeling unwell, muscles aches, headache, chills, rigors, nausea, fever, joint pain, urticaria/rash, and pruritus. Also information was collected if administration was slowed down or stopped for reactogenicity reasons.
Time Frame: About 30 minutes of product administration
Population: Subjects who received MAb114 (N=18), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: 5 mg/kg IV (n=3): Group 1 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 5 mg/kg.
  VRC-EBOMAB092-00-AB (MAb114): VRC-EBOMAB092-00-AB (MAb114) is a human immunoglobulin (IgG1) monoclonal antibody (MAb) targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP).
- Group 2: 25 mg/kg IV (n=5): Group 2 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 25 mg/kg.
  VRC-EBOMAB092-00-AB (MAb114): VRC-EBOMAB092-00-AB (MAb114) is a human immunoglobulin (IgG1) monoclonal antibody (MAb) targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP).
- Group 3: 50 mg/kg IV (n=10): Group 3 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 50 mg/kg.
  VRC-EBOMAB092-00-AB (MAb114): VRC-EBOMAB092-00-AB (MAb114) is a human immunoglobulin (IgG1) monoclonal antibody (MAb) targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP).
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=10)
Number analyzed (Participants) | 3 | 5 | 10
Participants
  Number who experienced infusion reaction | 0 | 0 | 0
  Number who completed infusion in about 30 min | 3 | 5 | 10

2. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 3 Days of Product Administration
Description: Subjects recorded 3-day systemic reactogenicity symptoms in a diary after study product administration. Solicited systemic symptoms include: unusually tired/feeling unwell, muscles aches, headache, chills, nausea, fever and joint pain. Subjects recorded highest measured temperature daily. Clinicians reviewed the diary with the subject and collected resolution information for any symptoms that were not resolved within 3 days. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects experiencing any systemic symptom as reported at the worst severity. Solicited reactogenicity was recorded without an attribution assessment. Grading was done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1.
Time Frame: 3 days after product administration
Population: Subjects who received MAb114 (N=18), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Overall (n=18): Total number of subjects who received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=10) | Overall (n=18)
Number analyzed (Participants) | 3 | 5 | 10 | 18
Participants
  Malaise: None | 3 | 4 | 8 | 15
  Malaise: Mild | 0 | 1 | 2 | 3
  Malaise: Moderate | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 4 | 9 | 16
  Myalgia: Mild | 0 | 1 | 1 | 2
  Myalgia: Moderate | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Headache: None | 3 | 3 | 8 | 14
  Headache: Mild | 0 | 2 | 2 | 4
  Headache: Moderate | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0
  Chills: None | 3 | 4 | 9 | 16
  Chills: Mild | 0 | 1 | 1 | 2
  Chills: Moderate | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Nausea: None | 3 | 4 | 9 | 16
  Nausea: Mild | 0 | 1 | 1 | 2
  Nausea: Moderate | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Fever: None | 3 | 5 | 10 | 18
  Fever: Mild | 0 | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0 | 0
  Joint Pain: None | 3 | 4 | 9 | 16
  Joint Pain: Mild | 0 | 1 | 1 | 2
  Joint Pain: Moderate | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0
  Any systemic symptom reported: None | 3 | 3 | 8 | 14
  Any systemic symptom reported: Mild | 0 | 2 | 2 | 4
  Any systemic symptom reported: Moderate | 0 | 0 | 0 | 0
  Any systemic symptom reported: Severe | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Product Administration
Description: Local reactogenicity symptoms were assessed and recorded by clinicians. Solicited local symptoms include pain/tenderness, swelling, redness, bruising, and pruritus (itchiness) at the product administration site. Clinicians assessed the study product administration site for local symptoms on the day of product administration after completion of the administration and on Days 1, 2 and 7 post administration. Subjects were counted once for each symptom at the worst severity if they experienced the symptom at any severity during the reporting period. If symptoms were experienced, clinicians collected resolution information for any symptom that wasn't resolved within 7 days. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom as reported at the worst severity. Solicited reactogenicity was recorded without attribution assessment. Grading was done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1.
Time Frame: 7 days after product administration
Population: Subjects who received MAb114 (N=18), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=10) | Overall (n=18)
Number analyzed (Participants) | 3 | 5 | 10 | 18
Participants
  Pain/Tenderness: None | 3 | 5 | 10 | 18
  Pain/Tenderness: Mild | 0 | 0 | 0 | 0
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0
  Bruising: None | 3 | 5 | 10 | 18
  Bruising: Mild | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0
  Swelling: None | 3 | 5 | 10 | 18
  Swelling: Mild | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0
  Redness: None | 3 | 5 | 10 | 18
  Redness: Mild | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0
  Pruritis: None | 3 | 5 | 10 | 18
  Pruritis: Mild | 0 | 0 | 0 | 0
  Pruritis: Moderate | 0 | 0 | 0 | 0
  Pruritis: Severe | 0 | 0 | 0 | 0
  Any Local Symptoms Reported: None | 3 | 5 | 10 | 18
  Any Local Symptoms Reported: Mild | 0 | 0 | 0 | 0
  Any Local Symptoms Reported: Moderate | 0 | 0 | 0 | 0
  Any Local Symptoms Reported: Severe | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects Reporting 1 or More Unsolicited Non-Serious Adverse Events
Description: Unsolicited adverse events (AEs) collected during the period from study product administration at Day 0 through 28 days after product administration. After the indicated time period through the last expected study visit at 24 weeks after product administration, only new chronic medical conditions collected as unsolicited AEs.
  The number reported is the number of subjects who experienced at least one AE in the reporting period. A subject with multiple experiences of the same event is counted once using the event of worst severity. The relationship between an AE and the product was assessed by the investigator on the basis of his or her clinical judgment and the protocol-specific definitions of Related - There is a reasonable possibility that the AE may be related to the study product and Not Related - There is not a reasonable possibility that the AE is related to the study product.
Time Frame: Through 24 weeks after product administration
Population: Subjects who received MAb114 (N=18), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=10) | Overall (n=18)
Number analyzed (Participants) | 3 | 5 | 10 | 18
Participants
  Related to MAb114 Administration | 0 | 0 | 0 | 0
  Not Related to MAb114 Administration | 0 | 2 | 5 | 7

5. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events (SAEs) collected during the period from study product administration at Day 0 through 24 weeks after product administration. Grading done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1. The relationship between a SAE and the product was assessed by the investigator on the basis of his or her clinical judgment and the protocol-specific definitions of Related - There is a reasonable possibility that the SAE may be related to the study product and Not Related - There is not a reasonable possibility that the SAE is related to the study product.
Time Frame: Through 24 weeks after product administration
Population: Subjects who received MAb114 (N=18), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=10) | Overall (n=18)
Number analyzed (Participants) | 3 | 5 | 10 | 18
Participants
  Related to MAb114 Administration | 0 | 0 | 0 | 0
  Not Related to MAb114 Administration | 0 | 0 | 1 | 1

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MAb114
Description: Cmax is the peak serum concentration that MAb114 achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-28 days post-infusion
Population: Subjects with 28 days of pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Group 3: 50 mg/kg IV (n=5): Group 3 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 50 mg/kg.
  VRC-EBOMAB092-00-AB (MAb114): VRC-EBOMAB092-00-AB (MAb114) is a human immunoglobulin (IgG1) monoclonal antibody (MAb) targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP).
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
µg/mL | 198.45 (45.15) | 829.38 (237.40) | 1961.21 (339.83)

7. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of MAb114
Description: Tmax is the time it takes to reach Cmax of MAb114 after it has been administered; it is determined based on the summary PK curve for each study group.
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-28 days post-infusion
Population: Subjects with 28 days of pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
hours | 3.21 (1.56) | 2.99 (2.16) | 2.75 (1.63)

8. Secondary Outcome: Mean Serum Concentration of MAb114
Description: The mean of individual subject MAb114 serum concentrations by administered dose group
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-28 days post-infusion
Population: Subjects with 28 days of pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
µg/mL
  Concentration at Day 7 | 52.60 (22.19) | 373.12 (75.32) | 692.64 (201.63)
  Concentration at Day 14 | 42.90 (5.53) | 272.91 (46.16) | 629.34 (118.19)
  Concentration at Day 28 | 25.46 (5.96) | 180.19 (38.82) | 427.21 (88.43)
  Average Concentration Days 0-28 | 52.87 (10.87) | 306.65 (32.14) | 663.87 (129.55)

9. Secondary Outcome: Overall IV Half-life (T1/2) of MAb114
Description: Half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-56 days post-infusion
Population: Subjects with 56 days of pharmacokinetic data. No standard deviation reported for a Group 3 single subject data.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Group 3: 50 mg/kg IV (n=1): Group 3 subjects received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0 at a dose of 50 mg/kg.
  VRC-EBOMAB092-00-AB (MAb114): VRC-EBOMAB092-00-AB (MAb114) is a human immunoglobulin (IgG1) monoclonal antibody (MAb) targeted to the Zaire ebolavirus (EBOV) glycoprotein (GP).
- Overall (n=9): Total number of subjects who received a single IV infusion of a Human Monoclonal Antibody (MAb), VRC-EBOMAB092-00-AB (MAb114), on Day 0
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=1) | Overall (n=9)
Number analyzed (Participants) | 3 | 5 | 1 | 9
days | 20.1 (6.9) | 26.7 (3.8) | 23.6 | 24.2 (1.8)

10. Secondary Outcome: Area Under the Curve (AUC0-28D)
Description: The AUC0-28D represents the total drug exposure in 28 days after MAb114 administration; it is determined based on the summary PK curve for each group.
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-28 days post-infusion
Population: Subjects with 28 days of pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: µg x day/mL
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
µg x day/mL | 1480 (304) | 8586 (900) | 18588 (3627)

11. Secondary Outcome: Volume of Distribution (Vd) at Steady-state
Description: Theoretical volume that would be necessary to contain the total amount of administered drug at the same concentration as observed in plasma. It represents the degree to which a drug is distributed in body tissue rather than the plasma and calculated based in the PK curve for each study group.
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-28 days post-infusion
Population: Subjects with 28 days of pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
Liters | 5.08 (0.88) | 3.93 (0.50) | 4.16 (0.74)

12. Secondary Outcome: MAb114 Clearance Rate
Description: Rate of MAb114 elimination divided by the plasma MAb114 concentration; determined based on the summary PK curve for each study group.
Time Frame: Pre-infusion (baseline), end of infusion (0h), 1 hr, 3 hr, 6 hr, 24 hr, 48 hr and 7-28 days post-infusion
Population: Subjects with 28 days of pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
mL/day | 199 (45) | 108 (21) | 115 (15)

13. Secondary Outcome: Number of Subjects Who Produced Anti-drug Antibodies to MAb114
Description: Serum samples collected 28 days and 56 days after MAb114 administration
Time Frame: Days 28 and 56 post-infusion
Population: Subjects with serum samples collected at 28 days and 56 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 5 mg/kg IV (n=3) | Group 2: 25 mg/kg IV (n=5) | Group 3: 50 mg/kg IV (n=5)
Number analyzed (Participants) | 3 | 5 | 5
Participants
  Day 28: Subjects with Anti-drug antibodies | 0 | 0 | 0
  Day 56: Subjects with Anti-drug antibodies: number analyzed (Participants) | 3 | 5 | 1
  Day 56: Subjects with Anti-drug antibodies | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) included systemic AEs reported by subjects at the worst severity through 3 days post product administration; and local administration site AEs reported at the worst severity through 7 days post product administration. Unsolicited AEs were reported from the date of product administration through 28 days thereafter, and new chronic medical conditions and SAEs with onset any time following the date of product administration through 24 weeks.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of subjects reporting the event. The total number of subjects affected in Other AEs includes subjects reporting at least one solicited and/or unsolicited AE. A subject with multiple experiences of the same event is counted once using the event of worst severity. Solicited events are reported separately from unsolicited events.
Arm/Group | Group 1: 5 mg/kg IV | Group 2: 25 mg/kg IV | Group 3: 50 mg/kg IV
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 1/10
Other Adverse Events (participants affected / at risk) | 0/3 | 3/5 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 5 mg/kg IV (N=3) | Group 2: 25 mg/kg IV (N=5) | Group 3: 50 mg/kg IV (N=10)
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 5 mg/kg IV (N=3) | Group 2: 25 mg/kg IV (N=5) | Group 3: 50 mg/kg IV (N=10)
Hordeolum (Infections and infestations) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Malaise (General disorders) | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 2
Chills (General disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03478891/Prot_SAP_ICF_002.pdf